CLINICAL TRIAL: NCT00538759
Title: RADiation Following Percutaneous Balloon Aortic Valvuloplasty to Prevent Restenosis
Acronym: RADAR
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Funding shortfall
Sponsor: Minneapolis Heart Institute Foundation (Other)
Collaborators: Twin Cities Heart Foundation (Unknown); Minneapolis Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: G060198
Record Dates: First submitted 2007-10-01; First posted 2007-10-03 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic valve stenosis; Balloon aortic valvuloplasty; Aortic valve restenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EBRT (Experimental): External beam radiation therapy to the aortic valve after successful balloon aortic valvuloplasty.
  Interventions: Device: External beam radiation therapy
- Control (Sham Comparator): Sham external beam radiation therapy to the aortic valve after successful balloon aortic valvuloplasty.
  Interventions: Other: Sham Control

INTERVENTIONS:
Device: External beam radiation therapy — Experimental beam radiation therapy to the aortic valve after successful balloon aortic valvuloplasty
  Arms: EBRT
Other: Sham Control
  Arms: Control

SUMMARY:
The objective of the RADAR trial is to determine the impact of External Beam Radiation Therapy (EBRT) on aortic valve restenosis following successful percutaneous balloon aortic valvuloplasty (BAV) in elderly patients with severe calcific aortic stenosis.

DETAILED DESCRIPTION:
The RADAR trial is a prospective, randomized, double-blind, sham-controlled, two-stage, adaptive clinical trial. Following successful Balloon Aortic Valvuloplasty, patients with severe aortic stenosis will be randomized in a 2:1 fashion to External Beam Radiation Therapy (EBRT) plus standard medical therapy or standard medical therapy along with sham EBRT (placebo). During Stage One, approximately 110 patients will be enrolled in order to have 80 patients randomized and 66 patients with valid 6 month data. The sample size for Stage Two will be calculated at the end of Stage One. At the time of study commencement, the expectation is that the total sample size will be approximately 155 patients with valid 6-month data, and thus 195 will be randomized and up to 250 enrolled.

Patients will be followed for a period of two (2) years. Echocardiographic and clinical endpoint data will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Calcific aortic valve stenosis with an echocardiographically derived AV index of less than 0.45 cm2/m2.
* Any symptoms of severe AS, including near syncope/syncope, angina, excessive fatigue and/or shortness of breath with NYHA functional class II-IV limitation.
* Age greater than 75 and risk of aortic valve replacement surgery greater than or equal to 15 percent. This may be assessed by using the STS Risk Predictor (see appendix C), confirmed by consultation with a cardiac surgeon experienced in high risk aortic valve surgery
* OR by having a cardiac surgeon experienced in high risk aortic valve surgery document comorbid conditions (such as porcelain aorta, malnutrition or other comorbidities not captured by the STS scoring system) that make the risk greater than or equal to 15 percent by the estimation of the surgeon.
* If age greater than or equal to 90 a cardiac surgeon experienced in high risk aortic valve surgery must document that BAV is a better option for the patient than aortic valve replacement surgery.
* Probable survival greater than 6 months after successful valvuloplasty.
* Patient is competent, willing to comply with follow-up, understands risks, benefits and alternatives and has signed the Informed Consent form.

Exclusion Criteria:

* Patient has undergone previous BAV or AVR.
* Patient is undergoing BAV as a bridge to AVR.
* 4 plus (severe) Aortic insufficiency by echocardiogram obtained prior to planned BAV procedure.
* Known congenital AV abnormality (e.g., bicuspid AV).
* ST Elevation Myocardial Infarction (STEMI) associated with CKMB greater than or equal to 3 times ULN or stroke less than or equal to 6 weeks prior to planned BAV procedure.
* Bacterial endocarditis less than or equal to 1 year prior to planned BAV procedure.
* Left ventricular ejection fraction less than 30% by preprocedural echocardiography.
* Baseline mean AV gradient less than 30 mm Hg by echocardiogram unless associated with a left ventricular ejection fraction of less than 40 per cent and true severe AS confirmed by dobutamine stress echocardiogram, i.e., AVA index less than or equal to 0.45cm2/m2 at peak dobutamine infusion. See Appendix D for suggested protocol.
* Patients who do not achieve successful BAV performed as a part of RADAR Trial: success being defined as an improvement in 4-24 hour post-valvuloplasty echocardiographically-derived AVA that is greater than 35 per cent over baseline and AVA greater than or equal to 0.7 cm2 and the absence of 4+ plus AI.
* Percutaneous Coronary Intervention with drug eluting stent placement less than or equal to 6 months prior to planned BAV procedure or bare metal stent placement/balloon angioplasty less than or equal to 8 weeks prior to planned BAV procedure.
* Cardiogenic shock, as defined by a consistent systolic blood pressure less than 80 mm Hg off vasopressors or less than 90 mm Hg on vasopressors.
* Patients requiring ventilator support less than or equal to 48 hours prior to planned BAV procedure.
* Creatinine greater than 2.2 mg/dL less than or equal to 48 hours prior to planned BAV procedure.
* Platelet count less than or equal to 100,000/mm3 less than or equal to 48 hours prior to planned BAV procedure.
* Hemoglobin less than or equal to 9.0 gm/dL less than or equal to 48 hours prior to planned BAV procedure.
* Known allergy/sensitivity to ASA.
* Known allergy/sensitivity to both clopidogrel and ticlopidine.
* Gastrointestinal bleed requiring transfusion less than or equal to 2 weeks prior to planned BAV procedure.
* Prior external beam radiation therapy to the chest that, in the judgment of the radiation oncologist, will compromise patient safety or interfere with the interpretation of the study results. This includes any prior radiation to the thoracic contents, except for radiation treatments for malignant or benign lesions of the skin.
* Untreated pneumonia or other systemic infection associated with fever greater than 38.5˚c or WBC count greater than 10,000 less than or equal to 72 hours prior to planned BAV procedure.
* Concomitant medical illness (for example, terminal malignancy) that in the opinion of the investigator is associated with reduced survival of less than 6 months.
* Major surgery less than or equal to 2 weeks prior to planned BAV procedure.
* Any illness or condition which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results.
* Involvement in any study of an investigational drug, device or procedure less than or equal to 30 days prior to planned BAV procedure.
* Previous enrollment in this study.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wes R Pedersen, MD, Principal Investigator — Minneapolis Heart Institute Foundation
Locations (2):
- United States (2):
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Lindner Clinical Trial Center, Cincinnati, Ohio

REFERENCES:
- [Background] Pedersen WR, Van Tassel RA, Pierce TA, Pence DM, Monyak DJ, Kim TH, Harris KM, Knickelbine T, Lesser JR, Madison JD, Mooney MR, Goldenberg IF, Longe TF, Poulose AK, Graham KJ, Nelson RR, Pritzker MR, Pagan-Carlo LA, Boisjolie CR, Zenovich AG, Schwartz RS. Radiation following percutaneous balloon aortic valvuloplasty to prevent restenosis (RADAR pilot trial). Catheter Cardiovasc Interv. 2006 Aug;68(2):183-92. doi: 10.1002/ccd.20818. PMID 16810699
- See also: Minneapolis Heart Institute Foundation — http://www.mplsheart.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EBRT | Control
Started | 13 | 8
Completed | 13 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EBRT | Control | Total
Number analyzed (Participants) | 13 | 8 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 84.8 (4.8) | 84.3 (4.6) | 84.6 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 3 | 2 | 5
Diabetes [Count of Participants; unit: Participants] | 3 | 4 | 7
Hypertension [Count of Participants; unit: Participants] | 12 | 8 | 20
Hyperlipidemia [Count of Participants; unit: Participants] | 9 | 7 | 16
History of MI [Count of Participants; unit: Participants] | 2 | 3 | 5
Severe MR/MS [Count of Participants; unit: Participants] | 0 | 1 | 1
Severe TR/TS [Count of Participants; unit: Participants] | 1 | 0 | 1
Exertional dyspnea [Count of Participants; unit: Participants] | 10 | 8 | 18
Excessive fatigue [Count of Participants; unit: Participants] | 6 | 3 | 9
Syncope [Count of Participants; unit: Participants] | 3 | 3 | 6
B-Type Natriuretic Peptide (BNP) [Mean (Standard Deviation); unit: pg/ml] | 545 (522) | 744 (972) | 620 (710)

OUTCOME MEASURES:

1. Primary Outcome: Aortic Valve Area as a Continuous Variable, Measured by Echocardiography
Time Frame: 6 months
Population: Study was halted early due to funding shortfall. Did not reach enrollment goal
Measure: Mean (Standard Error); unit: cm^2
Groups:
- Control: Sham external beam radiation therapy to the aortic valve after successful balloon aortic valvuloplasty.
  Sham Control
Arm/Group | EBRT | Control
Number analyzed (Participants) | 10 | 7
cm^2 | 0.64 (0.06) | 0.72 (0.07)

2. Primary Outcome: Incidence of Major External Beam Radiation Therapy-related Complications
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | EBRT | Control
Number analyzed (Participants) | 13 | 8
Participants | 0 | 0

3. Secondary Outcome: NYHA Improvement
Description: Improvement from pre-procedural NYHA class. Patients' heart failure were graded according to the severity of their symptoms. The New York Heart Association (NYHA) Functional Classification was used. It places patients in one of four categories based on how much they are limited during physical activity.
  I No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  II Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  III Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  IV Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | EBRT | Control
Number analyzed (Participants) | 11 | 5
Participants | 6 | 4

4. Secondary Outcome: CHF Rehospitalization
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | EBRT | Control
Number analyzed (Participants) | 13 | 8
Participants | 5 | 3

5. Secondary Outcome: Aortic Valve Reintervention
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | EBRT | Control
Number analyzed (Participants) | 13 | 8
Participants | 8 | 1

6. Secondary Outcome: Aortic Valve Area Late Loss Index
Description: The difference between the Aortic Valve Area at 6 months and the Aortic Valve Area post procedure indexed to the subject
Time Frame: 6 months
Population: Study was halted early due to funding shortfall. Did not reach enrollment goal
Measure: Mean (Standard Error); unit: cm^2
Arm/Group | EBRT | Control
Number analyzed (Participants) | 10 | 7
cm^2 | 78.8 (13.6) | 40.7 (16.2)

7. Secondary Outcome: Aortic Valve Mean Gradient
Time Frame: 6 months
Population: Study was halted early due to funding shortfall. Did not reach enrollment goal
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | EBRT | Control
Number analyzed (Participants) | 10 | 7
mmHg | 48.6 (3.9) | 39.8 (4.6)

ADVERSE EVENTS:
Time Frame: Adverse events were collected out to two years
Arm/Group | EBRT | Control
All-Cause Mortality (participants affected / at risk) | 8/13 | 3/8
Serious Adverse Events (participants affected / at risk) | 12/13 | 7/8
Other Adverse Events (participants affected / at risk) | 13/13 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EBRT (N=13) | Control (N=8)
Anemia (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Arrhythmia (Cardiac disorders) | 3 (3) | 2 (2)
Aortic Valve Replacement (Cardiac disorders) | 3 (3) | 0 (0)
Balloon Valvuloplasty (Cardiac disorders) | 0 (0) | 1 (1)
Bleed (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cancer (General disorders) | 1 (2) | 0 (0)
Congestive Heart Failure Exacerbation (Cardiac disorders) | 5 (10) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Fatigue/Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Hepatic Ischemia (Cardiac disorders) | 1 (1) | 0 (0)
Hypoglycemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Multi-system Organ Failure (General disorders) | 1 (1) | 0 (0)
Non-cardiac Chest Pain (General disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneaumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Right Lower Lung
Acute Renal Failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Respiratory/COPD (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Aortic Valve Restenosis (Cardiac disorders) | 3 (4) | 0 (0)
Vertebraplasty (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EBRT (N=13) | Control (N=8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 5 (6)
Edema (General disorders) | 7 (8) | 3 (4)
Fatigue/Weakness (General disorders) | 6 (9) | 4 (4)
Non-Cardiac Chest Pain (General disorders) | 4 (9) | 4 (6)
Abrasion (General disorders) | 1 (1) | 0 (0)
Aches (General disorders) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 4 (5) | 2 (2)
Arrhythmia (Cardiac disorders) | 3 (4) | 0 (0)
Atrial Enlargement (Cardiac disorders) | 1 (1) | 0 (0)
Bleed (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Bone Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cardiomegaly (Cardiac disorders) | 2 (2) | 0 (0)
Congestive Heart Failure (Cardiac disorders) | 2 (2) | 2 (3)
Constipation/Fecal Impaction (Gastrointestinal disorders) | 2 (2) | 1 (1)
Chest Pain/Angina (Cardiac disorders) | 3 (4) | 3 (4)
Cramping (General disorders) | 1 (1) | 0 (0)
Dehydration (General disorders) | 1 (1) | 0 (0)
Diaphoresis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dizzy/Lightheaded (General disorders) | 2 (4) | 2 (2)
Ecchmyosis (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Groin Pain (Renal and urinary disorders) | 2 (2) | 3 (3)
Headache (General disorders) | 1 (1) | 2 (4)
Heart Murmur (Cardiac disorders) | 1 (1) | 0 (0)
Ulcer (Gastrointestinal disorders) | 2 (2) | 1 (1)
Hematoma (Blood and lymphatic system disorders) | 4 (5) | 1 (1)
Hemoptysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hyperkalemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Hypertension (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Hypoglycemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Hypomagnesemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypotension (Blood and lymphatic system disorders) | 6 (6) | 1 (2)
Hypoxemia (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Inflamation (General disorders) | 1 (1) | 1 (1)
Knee Replacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Luekopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Mental Status Change (Psychiatric disorders) | 2 (2) | 0 (0)
Urinary Issues (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 4 (4) | 0 (0)
Orthostatic Hypotension (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (2) | 0 (0)
Pulmonary Embolism (Cardiac disorders) | 0 (0) | 1 (1)
Pacemaker Generator Change (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory/COPD (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 1 (1)
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperdense Renal Lesions (Renal and urinary disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Upset Stomach/Vomit (Gastrointestinal disorders) | 2 (4) | 1 (1)
Worsening Aortic Stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Decreased Motor Function (General disorders) | 0 (0) | 1 (1) — Right Hand

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No